CLINICAL TRIAL: NCT01293201
Title: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study Evaluating the Safety and Efficacy of STAHIST in Adult and Adolescent Subjects With a History of Seasonal Allergic Rhinitis
Brief Title: Trial of STAHIST in Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Magna Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 105781-3
Record Dates: First submitted 2011-02-08; First posted 2011-02-10 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-04

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: SAR; Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- STAHIST Investigational Medical Product (Experimental): STAHIST Tablet, dosed one tablet BID
  Interventions: Drug: STAHIST
- Placebo (Placebo Comparator): Placebo tablet, identical appearance to IMP, dosed one tablet BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: STAHIST — STAHIST dosed one tablet, BID
  Arms: STAHIST Investigational Medical Product
Drug: Placebo — Placebo identical in appearance to IMP, dosed one tablet BID
  Arms: Placebo

SUMMARY:
The overall development plan is to show that the combination of tried-and-proven decongestant/antihistamine ingredients (pseudoephedrine hydrochloride and chlorpheniramine maleate), plus a very small amount of belladonna alkaloids (.24 mg atropine sulfate) is a comprehensive, safe and effective B.I.D. drug treatment regimen, indicated for the relief of symptoms associated with seasonal allergic rhinitis in adults and children 12 years of age and older. Treated symptoms include nasal congestion, sneezing, rhinorrhea, itchy nose, itchy/watery eyes, and post nasal drip syndrome [reduction in tickly cough (acute or chronic), mucus in the back of the throat, sore throat, and hoarseness]. Considering the favorable safety and efficacy results of Phase 1 and Phase 2, the purpose of Phase 3 is to assess and compare the safety and efficacy of the study drug in a larger group comparatively with a placebo control group. Objectives: A) To report and compare total symptom scores (TSS) by SAR subjects rating the efficacy of STAHIST vs. placebo in relieving nasal congestion, rhinorrhea, nasal itching, sneezing, and post-nasal drip over the two-week study period. B) Report any side effects or adverse drug reactions and rate the severity of any incident. C) Compare and report each symptom score, total nasal symptom scores (TNSS), and post-nasal drip symptom scores (PND-S) between the two study arms.

DETAILED DESCRIPTION:
Phase 3 clinical trial will be conducted in conformance with Good Clinical Practices and is a multi-center, double-blind, randomized, placebo-controlled, parallel-group study evaluating the safety and efficacy of STAHIST (IMP) in 300 adult and adolescent subjects 12-60 years of age, of either sex or any race with a minimum 2-year history of seasonal allergic rhinitis (SAR) and a baseline minimum total symptom score (TSS) of not less than 8 on the S5 Subject Diary. Subjects will be treated twice daily with IMP or placebo for a period of two weeks. Subjects will visit the study site for at least 4 visits: screening, randomization/study inception, end-of-week one, final visit, and unscheduled visits as appropriate.

Run In (washout period): Subjects will be required to stop using oral nasal decongestants or first generation antihistamines for 48 hours, second generation antihistamines and Singulair for seven days, systemic corticosteroids for 30 days, and nasal or ocular corticosteroid medications for two weeks. Use of these drugs will also not be allowed during the study.

The first dose will be administered at the study site and subjects will be monitored on-site for one hour following dosing. There will be 24-hour on-call telephone access between physician/office staff and study subjects.

A Study Flow Chart will be used to facilitate trial management, record completed tasks as well as document their time of completion (See Study Flow Chart and Source Documents-Appendix D).

Safety evaluations will include monitoring of subject-reported AEs, measurement of vital signs, and assessment of safety laboratory data. Qualified independent, non-study administration individuals will be selected prior to the start of treatment for the purpose of safety monitoring.

300 subjects will be randomized. Assuming a screen failure test rate of approximately 33%, approximately 450 subjects will be screened.

At the conclusion of the study, the CSR will be prepared by the Sponsor, reviewed and approved by the Principal/Coordinator Investigator before submission.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females of any ethnic group between 12 and 60 years of age.
2. History of moderate to severe Seasonal Allergic Rhinitis (SAR) for at least two years.
3. Subjects' symptoms resulting from the irritation of sinus, nasal and upper respiratory tract tissues will include the five symptoms ("S5") that are the focus of this study: nasal congestion, rhinorrhea, nasal itching, sneezing, and post nasal drip. Subjects must have an average TSS baseline score of at least 8 on the S5 Subject Diary.
4. Prior to study drug administration, subjects' good health will be confirmed by medical history & physical examination, including pregnancy test (urine dip) before study inception.
5. Allergic hypersensitivity will be confirmed by the physician or well established patient medical history.
6. Subject's compliance with requisite run-in period for the individual will be confirmed by the investigator/designee.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Immunotherapy unless at stable maintenance dose.
3. Presence of a medical condition that might interfere with treatment evaluation or require a change in therapy including but not limited to high blood pressure or urinary retention problems.
4. Alcohol dependence.
5. Use of any other investigational drug in the previous month.
6. Subjects presenting with asthma requiring corticosteroid treatment.
7. Subjects with multiple drug allergies.
8. Subjects known to have an idiosyncratic reaction to any of the ingredients in IMP.
9. Subject who has used any investigational drugs within 30 days of the screening visit.
10. Subject who is participating in any other clinical study.
11. Subject who is unable to meet washout requirements.
12. Subject with clinically significant abnormal vital sign or laboratory value that precludes participation.
13. Subjects with any family relationship to Sponsor, Investigator, or staff of Sponsor or Investigator.
14. A URI within 4 weeks of study inception.
15. Subjects taking beta blockers or tri-cyclic antidepressants will not be allowed to participate in the study.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 290 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Total Symptom Scores (TSS) | Every 12 hours, two weeks trial duration
  To report and compare total symptom scores (TSS) by SAR subjects rating the efficacy of STAHIST vs. placebo in relieving nasal congestion, rhinorrhea, nasal itching, sneezing, and post-nasal drip over the two-week study period.

SECONDARY OUTCOMES:
Adverse Events (AEs) Assessment | Every 12 hours, two weeks study duration
  B) Report any side effects or adverse drug reactions and rate the severity of any incident.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Pollard, MD, Principal Investigator — Family Allergy and Asthma Research Institute
Locations (8):
- United States (8):
  - Clinical Research Atlanta, Stockbridge, Georgia
  - The South Bend Clinic, South Bend, Indiana
  - Family Allergy and Asthma Institute, Louisville, Kentucky
  - Family Allergy and Asthma, Somerset, Kentucky
  - New Horizons Clinical Research, Cincinnati, Ohio
  - National Allergy, Asthma & Urticaria Centers of Charleston, PA, Charleston, South Carolina
  - Pharmaceutical Research and Consulting, Inc, Dallas, Texas
  - Central Texas Health Research, New Braunfels, Texas